CLINICAL TRIAL: NCT05746858
Title: Deciphering the Biology of Relapsed/Refractory Diffuse Large B Cell Lymphoma (R/R DLBCL) Subtypes: Identification of Predictive Biomarkers Including miRNA-based Tumor Signatures to Optimize Sequential Treatment Decisions. (MIMOSA)
Brief Title: Predictive Biomarkers Including miRNA-based Tumor Signatures in Diffuse Large B Cell Lymphoma (R/R DLBCL) (MIMOSA)
Acronym: MIMOSA
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Istituti Fisioterapici Ospitalieri (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Sponsor
Other Study IDs: ID-5444
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Diffuse Large B Cell Lymphoma; Relapsed Non-Hodgkin Lymphoma
Keywords: miRNA; flow cytometry; next generation sequencing
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * Tissue samples in FFPE and fresh tissue samples
  * Plasma/serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention (observational study) — No intervention (observational study)

SUMMARY:
The goal of this study is to identify biomarkers that will predict outcome to standard and targeted therapies in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL). The specific aims of the present project are:

1. To explore associations between expression of target antigens on surface of neoplastic cells of DLBCL patients and response to target therapies
2. To identify specific miRNA signatures as predictors of response to upfront and salvage immune-chemotherapies in DLBCL patients.
3. To refine the diagnosis and molecular profiling of DLBCL, and to provide biological information of prognostic relevance in the setting of innovative treatments of patients with DLBCL.

DETAILED DESCRIPTION:
The research activities will be conducted within a project-specific retrospective/ prospective, multicenter, non-interventional study. The study is non-interventional since all patients will be treated according to institutional guidelines for standard clinical practice at each center.

Duration of the study: this is a two-year project, in the first 4 moths the retrospective part of the study will be performed, the accrual of patients for the prospective part will start rom the fourth month and the analysis of the prospective samples will last until the end of the project. The in vitro model will be established during the first year and the in vitro experiments will be performed until the enst of the project. The last months of the study will be dedicated to the statistical analysis of data and to their interpretation.

This project will be developed through the following specific Tasks:

Task 1: To explore associations between expression of target antigens on surface of neoplastic cells of DLBCL patients and response to target therapies A flow cytometric algorithm has been developed to identify an aberrant CD19+ B cell populations suggestive for aggressive B cell lymphoma that consists in the identification of a cell population defined by either the presence of surface immunoglobulin light chain clonality or the absence of light chains expression in combination with increased FSC and SSC physical parameters. These populations will be analysed for expressioe of target antigens.

Task 2: To identify specific miRNA signatures as predictors of response to upfront and salvage immunotherapies in DLBCL patients.

To this end miRNA expression profiling will be performed by Nanostring technology in formalin fixed and paraffin embedded (FFPE) tumor tissue samples collected at diagnosis. The resulting hits will be further analyzed in matched plasma/serum samples to evaluate the potential use of miRNAs as non-invasive biomarkers.

Task 3: To refine the diagnosis and molecular profiling of DLBCL, and to provide biological information of prognostic relevance in the setting of innovative treatments of patients with DLBCL The major aim is to provide the multilevel characterization (nanostring, NGS) of DLBCL cases that are concurrently utilized to develop a miRNA signature predictive of response to upfront and salvage treatments. Cases will be also characterized for structural alterations of MYC, BCL2 and BCL-6 genes (FISH) and for dual MYC/BCL2 protein expression (immunohistochemistry). In addition, information on pathways of immunosurveillance and microenvironmental functions will be generated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DLBCL and RR-DLBCL;
* Age>18 years;
* Eligibility for first-line and/or salvage chemo-immunotherapies as above specified;
* Measurable and/or evaluable disease (at least one bi-dimensionally measurable lesion on imaging scan defined as >1.5 cm in its longest dimension);
* No concomitant active cancers or others life-threatening conditions that can compromise chemotherapy treatment;
* Available FFPE and fresh tumor tissue (excisional biopsy, Tru-cut microhistology);
* Informed consent to treatment and use of biologic materials for studies related to the present proposal.

Exclusion Criteria:

* Diagnosis of follicular lymphoma grade 3b, lymphoblastic lymphoma, Burkitt lymphoma or primary mediastinal lymphoma;
* Age ≤ 18 years;
* Ineligible for first-line and/or salvage chemo-immunotherapies;
* No measurable and/or evaluable disease;
* Patients with concomitant active solid tumors or others clinical conditions that can compromise chemotherapy treatment or negatively influence the prognosis;
* Known history of HIV seropositive status. HIV testing will be performed at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a) newly diagnosed DLBCL patients treated with: i) standard R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone) and DA-EPOCH -R regimens; ii) frontline Pola-R-CHP (Polatuzumab vendotin, Rituximab, Cyclophosphamide, Doxorubicin, Prednisone) as approved by the European Medicine Agency-CHMP (24.03.2022); b) RR-DLBCL patients receiving salvage treatments including: a) R-Pola-Benda (Rituximab, Polatuzumab vendotin, Bendamustine); b) Lenalidomide-Tafasitamab; c) Anti-CD19 CAR-T cells; d) bispecific antibodies (e.g. Glofitamab).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 2 years
  Complete remission rates according to miRNA signatures, expression of target antigens, mutational status

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hohaus, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli
Locations (3):
- Italy (3):
  - Istituto Nazionale Tumori Fondazione "G. Pascale" IRCCS, Napoli
  - Fonadazione Policlinico Universitario A. Gemelli, Roma
  - Istituti Fisioterapici Ospitalieri -Istituto Regina Elena, Roma

IPD SHARING:
Plan to Share IPD: Undecided
Decision on IPD will be jointly made by investigators at end of study